CLINICAL TRIAL: NCT02470325
Title: A Randomized Double Blind Study of Cannabis on Dystonia and Spasticity in Pediatric Patients
Brief Title: The Effects of Cannabis on Dystonia and Spasticity on Pediatric Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Luba Blumkin, Dr. Luba Blumkin, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0101-14-WOMC
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Spasticity; Dystonia
Keywords: Cerebral palsy; Genetic neurodegenerative diseases
MeSH Terms: conditions — Muscle Spasticity; Dystonia; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 Avidekel (Active Comparator): Patients with spasticity and dystonia related to genetic neurodegenerative disease will consume Avidekel oil (6-to-1 ratio of CBD to THC)
  Interventions: Drug: Avidekel oil
- 2 Enriched Avidekel (Active Comparator): Patients with spasticity and dystonia related to genetic neurodegenerative disease will consume Enriched Avidekel oil (20-to-1 ratio of CBD to THC)
  Interventions: Drug: Enriched Avidekel oil
- 3 Avidekel (Active Comparator): Patients with spasticity and dystonia due to cerebral palsy will consume Avidekel oil (6-to-1 ratio of CBD to THC)
  Interventions: Drug: Avidekel oil
- 4 Enriched Avidekel (Active Comparator): Patients with spasticity and dystonia due to cerebral palsy will consume Enriched Avidekel oil (20-to-1 ratio of CBD to THC)
  Interventions: Drug: Enriched Avidekel oil

INTERVENTIONS:
Drug: Avidekel oil — Avidekel cannabis oil 6:1 CBD:THC
  Other Names: Avidekel cannabis oil
  Arms: 1 Avidekel; 3 Avidekel
Drug: Enriched Avidekel oil — Enriched Avidekel cannabis oil 20:1 CBD:THC
  Other Names: Enriched Avidekel cannabis oil
  Arms: 2 Enriched Avidekel; 4 Enriched Avidekel

SUMMARY:
A clinical trial is planned to study the effects of cannabis on dystonia and spasticity in children with neurological diseases. The clinical trial will include 40 children divided into two groups: children with spasticity and dystonia due to cerebral palsy, and children with spasticity and dystonia due to genetic neurodegenerative diseases. Each group will be randomly divided into two arms and will receive Avidekel cannabis oil 6-to-1 ratio of CBD to THC or enriched Avidekel cannabis oil 20-to-1 ratio of CBD to THC. During the study, various variables will be collected including: medication intake, spasticity, dystonia score, pain scale, restlessness scale, quality of life measures, safety tests, side effects, and an addiction test. The investigators hypothesize that cannabis consumption will reduce dystonia and spasticity in children with motor disability related to genetic neurodegenerative diseases and cerebral palsy and as a result improve motor function, non-motor functions and quality of life.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effect of two cannabis oils containing the main cannabinoid Δ9 -THC and CBD ratio of 1 to 6 and 1 to 20 (respectively), on spastic movement disorder and dystonia.

40 children will be enrolled in this study and will be divided into 2 groups:

1. Children with spasticity and dystonia due to cerebral palsy
2. Children with spasticity and dystonia due to genetic neurodegenerative diseases

Each group will be randomly divided into two groups:

I. Active comparator: 6-to-1 ratio of CBD to THC oil II. Active comparator: 20-to-1 ratio of CBD to THC oil

During the study the following variables will be collected:

* Consumption of drugs \ medication intake
* Spasticity grade measured using the Modified Ashworth Scale
* Dystonia grade measured using the Barry Albright Dystonia Scale
* Patient's subjective report about the severity of his/her spasticity and/or dystonia
* Pain scale
* Restlessness scale
* Quality of life measures: function, sleep, mood , appetite , weight
* Safety tests: liver function, renal function, blood tests (complete blood chemistry), blood pressure, pulse, ECG
* Side effects
* Addiction test

The purposes of the study:

1. Efficiency - examining the effect of cannabis on dystonia and spasticity.
2. Examining the most effective cannabinoid ratio for the relief of dystonia and spasticity. (Δ9 -THC and CBD ratio of 1 to 6 or 1 to 20, respectively).
3. Examining the effect of cannabis on quality of life measures (such as medication intake, mood, appetite, sleep).
4. Safety: examination of side effects and unwanted effects of cannabis and its limitations.

Research Hypothesis: The investigators hypothesize that cannabis consumption will reduce dystonia and spasticity symptoms in children with motor disability related to genetic neurodegenerative diseases and cerebral palsy and as a result improves motor function, non-motor function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children ages one to 18 years old with a diagnosis of cerebral palsy or motor disability; spastic in light of neurodegenerative disease
* Standard ECG test results and stable health condition

Exclusion Criteria:

* Participants that have been diagnosed with psychosis.
* Abnormal ECG test results

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changing in Spasticity and Dystonia grades using Modified Ashworth Scale, Barry Albright Dystonia Scale and Patient's subjective report | Approximately 2 years

SECONDARY OUTCOMES:
Quality Of Life Scores on the Visual Analog Scale and CPCHILD questionnaire | Approximately 2 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately 2 years
Comparing the scores receive from the different scales in both groups to determine the most effective cannabis oil - a ratio of 1 to 6 or 1 to 20 of Δ9 -THC to CBD. | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Lubov Blumkin, Holon, Israel, Israel